CLINICAL TRIAL: NCT06223698
Title: Optimizing Extended Adjuvant Endocrine Therapy in Patients With Breast Cancer: a Registry-based Randomized Clinical Trial - SWE-Switch Breast Cancer Trial
Brief Title: Optimizing Extended Adjuvant Endocrine Therapy in Patients With Breast Cancer
Acronym: SWE-Switch
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Mid-Sweden Regional Cancer Centre (Unknown); Akademiska University Hospital, Uppsala, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280050
Record Dates: First submitted 2023-12-29; First posted 2024-01-25 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant therapy; endocrine treatment; extended therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole; exemestane; Tamoxifen

STUDY DESIGN:
Intervention Model Description: Two separate cohorts will be randomized (two arms in each study cohort)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Aromatase inhibitors for 5 years (Experimental): Cohort 1 (premenopausal at diagnosis => postmenopausal at randomization) 5-year tamoxifen => Randomized to Arm A (switching to aromatase inhibitors for 5 years).
  Interventions: Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane
- Cohort 1: Tamoxifen for 5 years (Active Comparator): Cohort 1 (premenopausal at diagnosis => postmenopausal at randomization) 5-year tamoxifen => Randomized to Arm B (continuing with tamoxifen for 5 years).
  Interventions: Drug: Tamoxifen
- Cohort 2: Tamoxifen for 5 years (Experimental): Cohort 2 (postmenopausal at diagnosis) 5-year aromatase inhibitors => Randomized to Arm A (switching to tamoxifen for 5 years).
  Interventions: Drug: Tamoxifen
- Cohort 2: Aromatase inhibitors for 2 years (Active Comparator): Cohort 2 (postmenopausal at diagnosis) 5-year aromatase inhibitors => Randomized to Arm B (continuing with AI for 2 years).
  Interventions: Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg daily
  Arms: Cohort 1: Aromatase inhibitors for 5 years; Cohort 2: Aromatase inhibitors for 2 years
Drug: Anastrozole — Anastrozole 1 mg daily
  Arms: Cohort 1: Aromatase inhibitors for 5 years; Cohort 2: Aromatase inhibitors for 2 years
Drug: Exemestane — Exemestane 25 mg daily
  Arms: Cohort 1: Aromatase inhibitors for 5 years; Cohort 2: Aromatase inhibitors for 2 years
Drug: Tamoxifen — Tamoxifen 20 mg daily
  Arms: Cohort 1: Tamoxifen for 5 years; Cohort 2: Tamoxifen for 5 years

SUMMARY:
Based on the risk of late recurrence in breast cancer patients with luminal disease with high-risk for recurrence, extended adjuvant endocrine therapy beyond 5 years is recommended as a valid treatment option. In premenopausal women at diagnosis converted to postmenopausal after the first five years of tamoxifen, two treatment strategies for extended adjuvant endocrine therapy are available, namely continuing with tamoxifen or switching to aromatase inhibitors (AI). No randomized evidence does exist and both treatment strategies are used in clinical practice. In postmenopausal women with higher recurrence risk initially treated with AI for five years, extended adjuvant therapy with additional two years of AI has shown to be as effective as additional five years of AI. However, no randomized evidence on whether a switching strategy of five-year extended tamoxifen is better compared to two-year extended AI is available. Both treatment strategies are used in clinical practice.

The primary objective of this register-based randomized trial is to investigate the overall survival between patients treated with switching strategy for extended adjuvant endocrine therapy compared to continuing with the same treatment as the initial 5 years in two different clinical scenarios:

* In premenopausal women at diagnosis who converted to postmenopausal after 5 years of tamoxifen.
* In postmenopausal women at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (premenopausal women at diagnosis converted to postmenopausal)

1. Women who were pre- or perimenopausal at diagnosis
2. Luminal breast cancer (defined as estrogen-receptor positive >/=10%, HER2-negative disease).
3. Treated with tamoxifen for at least 80% of a 5-year period (+/- 6 months from treatment completion).
4. No clinical signs of metastasis after 5 years tamoxifen treatment.
5. cN+ breast cancer at diagnosis indicating the need for extended adjuvant endocrine therapy.
6. Postmenopausal status at study entry defined according to the National Comprehensive Cancer Network Guidelines.

Cohort 2 (postmenopausal women at breast cancer diagnosis)

1. Women who were postmenopausal at diagnosis.
2. Luminal breast cancer (defined as estrogen-receptor positive >/=10%, HER2-negative disease).
3. Treated with AI for at least 80% of a 5-year period (+/- 6 months from treatment completion).
4. No clinical signs of metastasis after 5 years AI treatment.
5. cN+ breast cancer at diagnosis indicating the need for extended adjuvant endocrine therapy.

Exclusion Criteria:

Cohort 1

1. Prior invasive breast cancer diagnosis.
2. Other invasive malignancy within 5 years before or after breast cancer diagnosis
3. Non-luminal breast cancer (defined as estrogen-receptor < 10%).
4. Patients who were unable to complete at least 80% of 5-year initial treatment with tamoxifen.
5. Uncertain menopausal status (unable to evaluate menopausal status according to aforementioned definitions).
6. Recurrent or metastatic breast cancer within or after 5-year initial treatment with tamoxifen (DCIS-only is allowed at any time before or after breast cancer diagnosis).

8) Unable to give informed consent in Swedish. Cohort 2

1. Prior invasive breast cancer diagnosis.
2. Other invasive malignancy within 5 years before or after breast cancer diagnosis; non-Luminal breast cancer (defined as estrogen-receptor < 10%).
3. Patients who were unable to complete at least 80% of 5-year initial treatment with AI.
4. Recurrent or metastatic breast cancer within or after 5-year initial treatment with AI (DCIS-only is allowed at any time before or after breast cancer diagnosis).

6) No contraindication for tamoxifen therapy. 7) Unable to give informed consent in Swedish.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3832 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2032-05-02 (Estimated); Study Completion 2035-05-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 120 months

SECONDARY OUTCOMES:
Invasive disease-free survival | 36 months; 60 months; 120 months
Distant disease-free survival | 36 months; 60 months; 120 months
Breast cancer-specific survival | 36 months; 60 months; 120 months
Overall survival | 36 months; 60 months
Frequency of selected grade 3/4 toxicities | 36 months; 60 months; 120 months
  Selected grade 3 or 4 toxicities that lead to hospitalization will be captured and analyzed for each study arm.
Overall quality of life (EORTC QLQC30) | 24 months; 60 months
  Assessment of overall quality of life through global health status from EORTC QLQC30 (scale 0 to 100; higher score indicates better overall quality of life)
Adherence to treatment strategies (medical possession ratio) | 36 months; 60 months; 120 months
  Adherence will be calculated by using medication possession ratio (MPR; the sum of the days' supply for all fills of a given drug in a particular time period, divided by the number of days in the time period). A MPR of >/= 80% is defined as good adherence
Duration of sick leave | 36 months; 60 months; 120 months

CONTACTS AND LOCATIONS:
Locations (15):
- Sweden (15):
  - Visby Hospital, Visby, Gotland County
  - General Hospital of Eskilstuna, Eskilstuna
  - Falun County Hospital, Falun
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Ryhov County Hospital, Jönköping
  - Kalmar Hospital, Kalmar
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - St Göran Capio Hospital, Stockholm
  - University Hospital of Umeå, Umeå
  - Akademiska University Hospital Uppsala, Uppsala
  - Växjö Hospital, Vaxjo
  - Västerås General Hospital, Västerås

IPD SHARING:
Plan to Share IPD: Undecided